CLINICAL TRIAL: NCT06764355
Title: Total Neoadjuvant Therapy With Induction Immunochemotherapy and Chemoradiotherapy Followed by Surgery for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Immunochemotherapy and Chemoradiotherapy Followed by Surgery for Advanced Esophageal Squamous Cell Carcinoma
Acronym: NICE-ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202409007MIPE
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: ESCC; Total Neoadjuvant Treatment; Pathological Complete Response
Keywords: ESCC
MeSH Terms: interventions — tislelizumab; Paclitaxel; Cisplatin; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Total Neoadjuvant Therapy (Experimental): "neoadjuvant immunochemotherapy" and "chemoradiotherapy"
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Chemoradiotherapy

INTERVENTIONS:
Drug: Tislelizumab — 200 mg, 1h-IVF, Q3W on day 1 for 2 cycles
Drug: Paclitaxel — Paclitaxel 175 mg/m2, 3h-IVF, Q3W on day 1 for 2 cycles
Drug: Cisplatin — Cisplatin 75 mg/m2, 2h-IVF, Q3W on day 1 for 2 cycles
Radiation: Chemoradiotherapy — Chemoradiotherapy
  * Paclitaxel 50 mg/m2, 1h-IVF, on days 1, 8,15, 22, and 29;
  * Cisplatin 30 mg/m2,1h-IVF, on days 1, 8,15, 22, and 29;
  * RT: 1.8 Gy/fraction, 5 days a week, for 25 fractions (total dose= 45 Gy).

SUMMARY:
Effective systemic therapy such as nivolumab as an adjuvant therapy has been demonstrated to improve the outcomes of patients receiving neoadjuvant chemoradiotherapy (CRT) for locoregional esophageal cancer. A more effective systemic therapy with anti-PD-1 or anti-PD-L1 immune checkpoint inhibitors (ICIs) plus cisplatin-based doublet chemotherapy, which has shown with high tumor response rate and improved survivals in patients with late-stage ESCC, may provide crucial benefit to patients with locally advanced disease by improving the systemic control, downstaging the locoregional tumor burden and reducing recurrence and metastasis.

Collectively, the investigators hypothesize that total neoadjuvant therapy (TNT) approach-consisting of induction immunochemotherapy followed by CRT-is a promising strategy to enhance the outcomes for participants with locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven squamous cell carcinoma of the intrathoracic esophagus.
2. Locally advanced disease, which is defined by the TNM system of the American Joint Committee on Cancer (AJCC) Cancer Staging System (8th edition), fulfilling one of the following criteria as determined by staging procedures (including but not limited to endoscopic ultrasound, computed tomography, bronchoscopy or positron emission tomography):

   1. cT3/4a, N0, M0;
   2. cT1-4a, N1-3, M0.
3. Tumor length longitudinal ≤ 10cm and radial ≤ 5cm.
4. The tumor must not extend more than 2cm into the stomach.
5. No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
6. Age ≥ 18 and ≤ 75 years old.
7. Performance status ECOG 0~1.
8. Adequate bone marrow reserves, defined as:

   1. white blood cells (WBC) ≥ 3,000/µl or neutrophil count (ANC) ≥ 1,500/µl;
   2. platelets ≥ 100,000/µl.
9. Adequate liver function reserves, defined as:

   1. hepatic transaminases ≤ 2.5 x upper limit of normal (ULN);
   2. serum total bilirubin ≤ 2.0 x upper limit of normal (ULN).
10. Adequate renal function: Creatinine ≤1.5 x upper normal limit or estimated creatinine clearance ≥ 50 ml/min (estimated by Cockcroft-Gault formulation)
11. Written informed consent.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be mandatory.
13. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Adenocarcinoma
2. Previous thoracic irradiation
3. Previous systemic chemotherapy
4. Has received prior therapy with an anti-PD-1 or anti-PD-L1
5. Synchronous diagnosis of squamous cell carcinoma in the aerodigestive tract, other than esophageal cancer.
6. Prior malignancy, except for the following:

   1. adequately treated basal cell or squamous cell skin cancer;
   2. in-situ cervical cancer;
   3. a "cured" malignancy more than 5 years prior to enrollment.
7. Significant co-morbid disease, which prohibits the conduction of immunochemotherapy, concurrent CRT, or radical surgery, such as active systemic infection, symptomatic cardiac or pulmonary disease, or psychiatric disorders.
8. Documented myocardial infarction within the 6 months preceding registration (pretreatment ECG evidence of infarct only will not exclude patients). Patients with a history of significant ventricular arrhythmia requiring medication. Patients with a history of 2nd or 3rd degree heart block.
9. Pre-existing motor or sensory neurotoxicity greater than grade 1.
10. Patients with prior allergic reactions to drug containing Cremophor, such as teniposide or cyclosporine.
11. Weight loss > 15%.
12. Dementia or altered mental status that would prohibit the understanding and completion of informed consent.
13. Estimated life expectancy less than 3 months.
14. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
15. Has a known history of active TB (Bacillus Tuberculosis)
16. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. Has known history of, or any evidence of active, non-infectious pneumonitis, interstitial lung disease or pulmonary fibrosis.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Patients with untreated chronic HBV or chronic HBV carriers whose HBV DNA is ≥500 IU/mL, or patients with active HCV. Patients who are inactive carriers or with treated and stable hepatitis B (detectable B surface antigen and HBV DNA <500 IU/mL); patients with non-reactive HCV can be enrolled. Patients with chronic HBV infection need to be treated with anti-HBV agents while receiving immunochemotherapy and chemoradiotherapy according to the local and institutional guidelines.
21. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.
22. Has received organ transplantation.
23. Has declined esophagectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | through study completion, an average of 6 months
  To evaluate the pathological complete response (pCR) rate of participants receiving total neoadjuvant therapy with induction immunochemotherapy and chemoradiotherapy (CRT) followed by surgery in operable ESCC.

SECONDARY OUTCOMES:
Major pathological response | through study completion, an average of 6 months
  defined as number of participants with residual tumor cells ≤10% at the time of surgery divided by the number of participants received esophagectomy
R0 resection rate | through study completion, an average of 6 months
  defined as number of participants with no gross residual disease, plus negative section margins (i.e., proximal, distal, and circumferential margins are all > 1 mm) according to pathological examination of esophagectomy specimen.
Disease-free survival | from esophagectomy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 50 months
  defined as the time from esophagectomy until evidence of disease recurrence or death in participants received esophagectomy.
Event-free survival | from enrollment to an event which may include radiographic progression, clinical progression, local or distant recurrence, second aerodigestive tract squamous cell carcinoma, and death from any cause, whichever came first, assessed up to 50 months
  defined as the time from enrollment to an event which may include radiographic progression, clinical progression, local or distant recurrence, second aerodigestive tract squamous cell carcinoma, and death.
Distant metastasis-free survival | from esophagectomy until evidence of distant metastasis recurrence or death from any cause, whichever came first, assessed up to 50 months
  defined as the time from esophagectomy until evidence of distant metastasis recurrence or death.
Overall survival | the time from enrollment to death from any cause, whichever came first, assessed up to 50 months
  defined as the time from enrollment to death.
Loco-regional recurrence rate | from esophagectomy until evidence of loco-regional metastasis recurrence or death from any cause, whichever came first, assessed up to 50 months
  defined as number of participants with loco-regional recurrence divided by the number of participants received esophagectomy
Distant metastasis rate | from esophagectomy until evidence of distant metastasis or death from any cause, whichever came first, assessed up to 50 months
  defined as number of participants with distant recurrence divided by the number of participants received esophagectomy

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No